CLINICAL TRIAL: NCT06945653
Title: An Assessment of Diversity, Equity and Inclusion Education in Anesthesiology: A Survey of the American Society of Anesthesiologists (ASA) Members
Brief Title: DEI Education in Anesthesiology
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0329
Record Dates: First submitted 2025-04-11; First posted 2025-04-25 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-03

CONDITIONS: Diversity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- American Society of Anesthesiologists Members: Current members of the American Society of Anesthesiologists. Members include learners at all levels - medical students, residents and fellows - as well as attending anesthesiologists, CRNAs, research staff, etc.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — The survey questions are aimed to assess the current state of diversity training in anesthesiology education. This survey serves as a needs assessment and will help gather information on the current state of DEI education within the specialty.

SUMMARY:
To date, there has not been an assessment of ASA members to determine satisfaction with DEI and cultural humility/structural competency education within institutions and programs. We developed a 24-question survey that will be distributed via email to current members of the American Society of Anesthesiologists. Members include learners at all levels - medical students, residents and fellows - as well as attending anesthesiologists, CRNAs, research staff etc. The survey questions are aimed to assess the current state of diversity training in anesthesiology education. This survey serves as a needs assessment and will help gather information on the current state of DEI education within the specialty. The results of the survey will serve as an impetus for improvement in this domain by developing novel educational modules and workshops on these topics, at the institutional level and nationwide.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist Member

Exclusion Criteria:

* Not a member of the American Society of Anesthesiologists

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Members of the American Society of Anesthesiologists, including learners at all levels - medical students, residents and fellows - as well as attending anesthesiologists, CRNAs, research staff, etc.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Demographic Characteristics | Through study completion, about 2 months
  Examine demographic characteristics such as gender, race, ethnicity distribution and practice settings of ASA members.
Current Knowledge | Through study completion, about 2 months
  Evaluate current knowledge of ASA members regarding DEI and structural competence. Questions will ask members about their familiarity with terms related to DEI and structural competence and if they believe it is important for these terms to be taught.
Training Methods | Through study completion, about 2 months
  Examine the distinct DEI, cultural competency/humility training methods at the program/institutional level as well as ASA member satisfaction with this education. Questions will ask members how much training they received, when they received training, what kind of training they received, and how satisfied they are with the training received.

IPD SHARING:
Plan to Share IPD: Undecided